CLINICAL TRIAL: NCT03876743
Title: How Many Opiates Should we Prescribe for Pain in Patients Undergoing Knee Arthroscopies and ACL Reconstructions?
Brief Title: Opiates Prescribing for Knee Arthroscopies and ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Vehniah Tjong, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STU00206152
Record Dates: First submitted 2018-03-20; First posted 2019-03-15 (Actual); Results first posted 2020-09-16 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Knee Injuries; ACL Injury
MeSH Terms: conditions — Knee Injuries; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1-Knee Arthroscopy (Experimental): Will have all of their post-operative prescriptions sent down to the pharmacy on the day of surgery to be collected.
  Interventions: Other: Group 1-Knee Arthroscopy
- Group 2-Knee Arthroscopy (Experimental): Will have all prescriptions sent to pharmacy with the exception of an opiate prescription. Instead, they will be handed a physical paper prescription. They will be instructed to only fill the prescription if absolutely needed.
  Interventions: Other: Group 2-Knee Arthroscopy
- Group 1-ACL reconstruction (Experimental): Will be prescribed 60 opiate tablets in addition to other routine post-operative pain medication regimens.
  Interventions: Other: Group 1-ACL reconstruction
- Group 2-ACL reconstruction (Experimental): Will be prescribed 30 opiate tablets in addition to other routine post-operative pain medication regimens.
  Interventions: Other: Group 2-ACL reconstruction

INTERVENTIONS:
Other: Group 1-Knee Arthroscopy — Will have all of their post-operative prescriptions sent down to the pharmacy on the day of surgery to be collected.
  Arms: Group 1-Knee Arthroscopy
Other: Group 2-Knee Arthroscopy — Will have all prescriptions sent to pharmacy with the exception of an opiate prescription. Instead, they will be handed a physical paper prescription. They will be instructed to only fill the prescription if absolutely needed.
  Arms: Group 2-Knee Arthroscopy
Other: Group 1-ACL reconstruction — Will be prescribed 60 opiate tablets in addition to other routine post-operative pain medication regimens.
  Arms: Group 1-ACL reconstruction
Other: Group 2-ACL reconstruction — Will be prescribed 30 opiate tablets in addition to other routine post-operative pain medication regimens.
  Arms: Group 2-ACL reconstruction

SUMMARY:
The purpose of the study is to determine if opiates are required to achieve adequate analgesia after knee arthroscopy and ACL reconstruction in outpatient surgery.

The investigators hypothesize that patients are frequently prescribed more opiates than are needed after surgery, resulting in excess medications that are at risk for misuse, diversion and contribution to the opioid epidemic.

DETAILED DESCRIPTION:
Perioperative pain management is an important aspect of quality patient care. Opioid pain medications are increasingly being used for pain control, with the United States writing over 250 million prescriptions for painkillers per year. Increased usage has led to unintended negative consequences for individuals and society. It is estimated that 46 people die each day from an overdose of prescription painkillers, and individual use can lead to the development of tolerance and worse treatment outcomes. Further issues arise when opioids are misused, it is estimated that non-therapeutic use has increased three fold in recent years. In the United States alone in 2006 the estimated total cost of opioid prescription misuse was $53.4 billion, of which $42 billion was attributed to lost productivity, $8.2 billion to criminal justice cost and the remainder drug abuse treatment and medical complications. The federal government has recognized this epidemic and raised a call for clinicians to more responsibly prescribe opiate pain medications.

Opiate use has increased in recent years, from 2000-2010 the use of opiates in office based visits nearly doubled from 11.3% to 19.6% whereas there was no change in the prescribing of non-opioid pharmacotherapies. Further, when specifically looking at new musculoskeletal pain visits, one half resulted in pharmacologic treatment, with the prescribing of non-opioid pharmacotherapies decreasing from 38% to 29% from 2000 to 2010, respectively. The clinical use of opioids for post-operative pain control has also been linked to the opioid epidemic and risk of future abuse. Legitimate opioid use before high school graduation is independently associated with a 33% increased risk of future misuse after high school.

It has been estimated that orthopedic surgeons prescribe 7.7% of all opioids in the United States.Special attention needs to be paid to the amount of opioid pain medications orthopedic surgeons prescribe to patients after ambulatory surgery, there is considerable variability among surgeon and procedure in regards to the amount of opioids to prescribe with many patients left with excess unused medication.An analysis of 250 patients undergoing outpatient upper extremity surgery found that on average patients consumed 10 opioid pills, with 19 pills left over and a total of 4,639 pills going unused in the cohort. Leftover prescription opioids are at risk for diversion to family and friends for nonmedical use. Further studies are needed to quantify the amount of opioids to prescribe for specific orthopedic procedures to limit excess narcotic use, misuse, diversion and contribution to the opioid epidemic.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to Northwestern Memorial Hospital (NMH) or to a Northwestern orthopaedic surgery faculty member's clinic undergoing knee arthroscopy with meniscus repair and/or debridement
* 18 years old or greater
* Ability to read and speak English

Exclusion Criteria:

* Revision surgery
* Oncologic surgery
* Arthroscopic knee surgery that involves procedures other than ACL or the meniscus (i.e PCL, LCL, MPFL)
* Patients currently taking narcotics, chronic pain management patients, history of substance abuse
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Patients currently taking narcotics, chronic pain management patients, history of substance abuse

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-07-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Medicine Department of Orthopaedic Surgery, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hartwell MJ, Selley RS, Terry MA, Tjong VK. Can We Eliminate Opioid Medications for Postoperative Pain Control? A Prospective, Surgeon-Blinded, Randomized Controlled Trial in Knee Arthroscopic Surgery. Am J Sports Med. 2020 Sep;48(11):2711-2717. doi: 10.1177/0363546520941861. Epub 2020 Aug 5. PMID 32755488

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 (Filled)-Knee Arthroscopy: Will have all of their post-operative prescriptions sent down to the pharmacy on the day of surgery to be collected.
  Group 1-Knee Arthroscopy: Will have all of their post-operative prescriptions sent down to the pharmacy on the day of surgery to be collected.
- Group 2 (as Needed)-Knee Arthroscopy: Will have all prescriptions sent to pharmacy with the exception of an opiate prescription. Instead, they will be handed a physical paper prescription. They will be instructed to only fill the prescription if absolutely needed.
  Group 2-Knee Arthroscopy: Will have all prescriptions sent to pharmacy with the exception of an opiate prescription. Instead, they will be handed a physical paper prescription. They will be instructed to only fill the prescription if absolutely needed.
- Group 1 (60)-ACL Reconstruction: Will be prescribed 60 opiate tablets in addition to other routine post-operative pain medication regimens.
  Group 1-ACL reconstruction: Will be prescribed 60 opiate tablets in addition to other routine post-operative pain medication regimens.
- Group 2(30)-ACL Reconstruction: Will be prescribed 30 opiate tablets in addition to other routine post-operative pain medication regimens.
  Group 2-ACL reconstruction: Will be prescribed 30 opiate tablets in addition to other routine post-operative pain medication regimens.
Period: Overall Study
Arm/Group | Group 1 (Filled)-Knee Arthroscopy | Group 2 (as Needed)-Knee Arthroscopy | Group 1 (60)-ACL Reconstruction | Group 2(30)-ACL Reconstruction
Started | 54 | 51 | 46 | 50
Completed | 48 | 47 | 42 | 43
Not Completed | 6 | 4 | 4 | 7
Not completed — Lost to Follow-up | 6 | 4 | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Group 2 (30)-ACL Reconstruction: Will be prescribed 30 opiate tablets in addition to other routine post-operative pain medication regimens.
  Group 2-ACL reconstruction: Will be prescribed 30 opiate tablets in addition to other routine post-operative pain medication regimens.
- Total: Total of all reporting groups
Arm/Group | Group 1 (Filled)-Knee Arthroscopy | Group 2 (as Needed)-Knee Arthroscopy | Group 1 (60)-ACL Reconstruction | Group 2 (30)-ACL Reconstruction | Total
Number analyzed (Participants) | 54 | 51 | 46 | 50 | 201
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 53 | 51 | 46 | 50 | 200
  >=65 years | 1 | 0 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.8 (12.5) | 43.2 (13.2) | 33.2 (8.9) | 31.3 (10.0) | 38.1 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 20 | 22 | 23 | 96
  Male | 23 | 31 | 24 | 27 | 105
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.2 (7.6) | 29.8 (7.9) | 26.4 (4.1) | 28.1 (6.0) | 28.4 (6.7)
Are you an active smoker? [Count of Participants; unit: Participants]
  Yes | 5 | 7 | 1 | 4 | 17
  No | 49 | 44 | 45 | 46 | 184
If no, have you ever consistently smoked cigarettes (daily for >1 month)? [Count of Participants; unit: Participants] — Population: Among participants who are not current smokers
  Participants
    number analyzed (Participants) | 49 | 44 | 45 | 46 | 184
    Yes | 2 | 7 | 4 | 2 | 15
    No | 47 | 37 | 41 | 44 | 169
What is your employment status? [Count of Participants; unit: Participants]
  Employed | 48 | 40 | 39 | 36 | 163
  Unemployed | 2 | 6 | 6 | 12 | 26
  Disabled | 1 | 2 | 0 | 1 | 4
  Retired | 3 | 3 | 1 | 1 | 8
Is this injury part of a workers compensation claim? [Count of Participants; unit: Participants]
  Yes | 0 | 1 | 1 | 1 | 3
  No | 54 | 50 | 45 | 49 | 198
Are you actively participating in sporting activities? [Count of Participants; unit: Participants]
  Yes | 14 | 16 | 26 | 32 | 88
  No | 40 | 35 | 20 | 18 | 113
At what level (i.e. professional, collegiate, recreational)? [Count of Participants; unit: Participants]
  Professional | 0 | 0 | 0 | 2 | 2
  Collegiate | 2 | 3 | 3 | 2 | 10
  Recreational | 12 | 13 | 25 | 29 | 79
  N/A | 40 | 35 | 18 | 17 | 110
Are you currently using narcotic pain medications (ex. Norco, Vicodin, Oxycontin/Oxycodone) ? [Count of Participants; unit: Participants]
  Yes | 0 | 0 | 0 | 0 | 0
  No | 54 | 51 | 46 | 50 | 201
Do you have a personal history of illicit substance abuse? [Count of Participants; unit: Participants]
  Yes | 0 | 0 | 0 | 0 | 0
  No | 54 | 51 | 46 | 50 | 201
Do you have a family history of illicit substance abuse? [Count of Participants; unit: Participants]
  Yes | 4 | 4 | 7 | 6 | 21
  No | 50 | 47 | 39 | 44 | 180
What is the highest level of education you have attained? [Count of Participants; unit: Participants]
  Completed High School | 12 | 7 | 6 | 11 | 36
  Undergraduate | 25 | 26 | 24 | 29 | 104
  Graduate | 17 | 18 | 16 | 10 | 61
What is your average yearly household income? [Count of Participants; unit: Participants]
  Less than $20,000 | 2 | 6 | 4 | 4 | 16
  $20,000 -$34,999 | 3 | 1 | 1 | 2 | 7
  $35,000 -$49,999 | 10 | 4 | 4 | 8 | 26
  $50,000 -$74,999 | 8 | 10 | 11 | 13 | 42
  $75,000 - $99,999 | 8 | 8 | 7 | 9 | 32
  $100,000 -$149,999 | 4 | 11 | 8 | 8 | 31
  $150,000 - $199,999 | 9 | 1 | 3 | 2 | 15
  $200,000 or more | 10 | 10 | 8 | 4 | 32

OUTCOME MEASURES:

1. Primary Outcome: Numeric Pain Rating Scale (NPRS) Pain Score
Description: 2 hours post-op; minimum score: 0 = no pain, maximum score: 10 = worst imaginable pain; lower value is better
Time Frame: 2 hours post-op
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1-Knee Arthroscopy | Group 2-Knee Arthroscopy | Group 1-ACL Reconstruction | Group 2-ACL Reconstruction
Number analyzed (Participants) | 48 | 47 | 43 | 42
score on a scale | 5.2 (1.8) | 5.3 (2.2) | 5.0 (2.7) | 5.6 (2.2)

2. Primary Outcome: Opiate Count
Description: 24 hours post-op
Time Frame: 24 hours post-op
Measure: Mean (Standard Deviation); unit: pills
Arm/Group | Group 1-Knee Arthroscopy | Group 2-Knee Arthroscopy | Group 1-ACL Reconstruction | Group 2-ACL Reconstruction
Number analyzed (Participants) | 48 | 47 | 43 | 42
pills | 1.4 (1.8) | 1.6 (1.6) | 2.5 (2.2) | 3.6 (2.4)

3. Primary Outcome: Side Effects, 24 Hours Post-op
Description: Number of Participants with Side Effects, 24 hours post-op
Time Frame: 24 hours post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1-Knee Arthroscopy | Group 2-Knee Arthroscopy | Group 1-ACL Reconstruction | Group 2-ACL Reconstruction
Number analyzed (Participants) | 48 | 47 | 43 | 42
Participants | 7 | 5 | 23 | 24

4. Primary Outcome: Numeric Pain Rating Scale (NPRS) Pain Scores
Description: 48 hours post-op; minimum score: 0 = no pain, maximum score: 10 = worst imaginable pain; lower value is better
Time Frame: 48 hours post-op
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1-Knee Arthroscopy | Group 2-Knee Arthroscopy | Group 1-ACL Reconstruction | Group 2-ACL Reconstruction
Number analyzed (Participants) | 48 | 47 | 43 | 42
score on a scale | 3.0 (2.1) | 3.5 (.4) | 4.2 (2.2) | 4.6 (2.2)

5. Primary Outcome: Opiate Count
Description: 48 hours post-op
Time Frame: 48 hours post-op
Measure: Mean (Standard Deviation); unit: pills
Arm/Group | Group 1-Knee Arthroscopy | Group 2-Knee Arthroscopy | Group 1-ACL Reconstruction | Group 2-ACL Reconstruction
Number analyzed (Participants) | 48 | 47 | 43 | 42
pills | 2.1 (2.8) | 2.5 (2.8) | 4.8 (4.4) | 6.0 (3.9)

6. Primary Outcome: Side Effects
Description: 48 hours post-op
Time Frame: 48 hours post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1-Knee Arthroscopy | Group 2-Knee Arthroscopy | Group 1-ACL Reconstruction | Group 2-ACL Reconstruction
Number analyzed (Participants) | 48 | 47 | 43 | 42
Participants | 7 | 5 | 24 | 25

7. Primary Outcome: Numeric Pain Rating Scale (NPRS) Pain Scores
Description: 7 days post-op; minimum score: 0 = no pain, maximum score: 10 = worst imaginable pain; lower value is better
Time Frame: 7 days post-op
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1-Knee Arthroscopy | Group 2-Knee Arthroscopy | Group 1-ACL Reconstruction | Group 2-ACL Reconstruction
Number analyzed (Participants) | 48 | 47 | 43 | 42
score on a scale | 2.0 (1.8) | 2.4 (2.3) | 2.9 (2.0) | 2.6 (1.8)

8. Primary Outcome: Opiate Count
Description: Number Pills Taken
Time Frame: 7 days post-op
Measure: Mean (Standard Deviation); unit: Pills Hydrocodone/Acetaminophen 10/325mg
Arm/Group | Group 1-Knee Arthroscopy | Group 2-Knee Arthroscopy | Group 1-ACL Reconstruction | Group 2-ACL Reconstruction
Number analyzed (Participants) | 48 | 47 | 43 | 42
Pills Hydrocodone/Acetaminophen 10/325mg | 3.5 (6.3) | 4.5 (6.0) | 9.5 (10.0) | 12.2 (14.2)

9. Primary Outcome: Number of Participants With Side Effects
Description: Potential side effects included lightheadedness, nausea, drowsiness, gastrointestinal symptoms, constipation
Time Frame: 7 days post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1-Knee Arthroscopy | Group 2-Knee Arthroscopy | Group 1-ACL Reconstruction | Group 2-ACL Reconstruction
Number analyzed (Participants) | 48 | 47 | 43 | 42
Participants | 7 | 5 | 24 | 25

10. Primary Outcome: Refill Requests
Description: Number of participants requesting opioid refills within 3 months after surgery
Time Frame: Within 3 months after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1-Knee Arthroscopy | Group 2-Knee Arthroscopy | Group 1-ACL Reconstruction | Group 2-ACL Reconstruction
Number analyzed (Participants) | 48 | 47 | 43 | 42
Participants | 1 | 0 | 5 | 7

11. Primary Outcome: Still Taking Opiates?
Description: Number of patients who took any opiates between surgery and 1 day postoperative
Time Frame: 1 day postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Filled)-Knee Arthroscopy | Group 2 (as Needed)-Knee Arthroscopy | Group 1 (60)-ACL Reconstruction | Group 2(30)-ACL Reconstruction
Number analyzed (Participants) | 48 | 47 | 43 | 42
Participants
  Yes | 38 | 30 | 38 | 39
  No | 10 | 17 | 5 | 3

12. Primary Outcome: Still Taking Opiates?
Description: Number of patients who took any opiates between 1 day and 2 days postoperative
Time Frame: 2 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Filled)-Knee Arthroscopy | Group 2 (as Needed)-Knee Arthroscopy | Group 1 (60)-ACL Reconstruction | Group 2(30)-ACL Reconstruction
Number analyzed (Participants) | 48 | 47 | 43 | 42
Participants
  Yes | 25 | 19 | 33 | 33
  No | 23 | 28 | 10 | 9

13. Primary Outcome: Still Taking Opiates?
Description: Number of patients who took any opiates between 2 days and 7 days postoperative
Time Frame: 7 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Filled)-Knee Arthroscopy | Group 2 (as Needed)-Knee Arthroscopy | Group 1 (60)-ACL Reconstruction | Group 2(30)-ACL Reconstruction
Number analyzed (Participants) | 48 | 47 | 43 | 42
Participants
  Yes | 18 | 17 | 29 | 31
  No | 30 | 30 | 14 | 11

14. Primary Outcome: Still Taking Opiates?
Description: Number of patients who took any opiates between 7 days and 21 days postoperative
Time Frame: 21 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Filled)-Knee Arthroscopy | Group 2 (as Needed)-Knee Arthroscopy | Group 1 (60)-ACL Reconstruction | Group 2(30)-ACL Reconstruction
Number analyzed (Participants) | 48 | 47 | 43 | 42
Participants
  Yes | 3 | 0 | 5 | 5
  No | 45 | 47 | 38 | 37

ADVERSE EVENTS:
Time Frame: 21 days post-surgery
Arm/Group | Group 1-Knee Arthroscopy | Group 2-Knee Arthroscopy | Group 1-ACL Reconstruction | Group 2-ACL Reconstruction
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/47 | 0/43 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/47 | 0/43 | 0/42
Other Adverse Events (participants affected / at risk) | 0/48 | 0/47 | 0/43 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/43/NCT03876743/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT03876743/SAP_001.pdf